CLINICAL TRIAL: NCT01600339
Title: A Single Arm, Multicenter, Open-label Phase II Trial of Cabazitaxel as Second Line Treatment of Patients With Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: A Trial of Cabazitaxel for Advanced Transitional Cell Carcinoma (TCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISGUOG1101.CTIL
Record Dates: First submitted 2012-02-26; First posted 2012-05-17 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CABAZITAXEL (Experimental): cabazitaxel at a starting dose of 25 mg/m
  Interventions: Drug: CABAZITAXEL

INTERVENTIONS:
Drug: CABAZITAXEL — The patients are planned to receive cabazitaxel at a starting dose of 25 mg/m(2) intravenously over 1 h, following premedication as accepted with cabazitaxel. Treatment cycles are every 3 weeks. All patients will receive primary GCSF support.

SUMMARY:
In this phase II multicenter study, the investigators aim to evaluate the efficacy and tolerability of a novel taxane-cabazitaxel as single agent second-line chemotherapy for metastatic urothelial carcinoma.

DETAILED DESCRIPTION:
For those patients with advanced bladder cancer who have progressed on a platinum based regimen, no widely accepted standard second line therapy currently exists. Taxanes including paclitaxel and docetaxel have exhibited limited clinical activity in this disease and are sometimes given off study. Cabazitaxel is a novel semi-synthetic taxane with a low affinity for the multidrug resistance 1 protein. In cell lines cabazitaxel is as potent as docetaxel, but in tumor cells that are resistant to taxanes, cabazitaxel overcome taxanes resistance.

In recent clinical data, this drug was shown to have potent activity in patients with metastatic prostate cancer resistant to docetaxel. Based on this phase III data, cabazitaxel was recently approved in the US, Europe and in Israel for these patients. The main toxicity of this taxane is neutropenia and diarrhea, thus primary prevention with GCSF may reduce the main toxicity of this agent.

In this phase II multicenter study, the investigators aim to evaluate the efficacy and tolerability of this novel taxane -cabazitaxel as single agent second-line chemotherapy for metastatic urothelial carcinoma after failure of prior platinum-based chemotherapy.

The patients are planned to receive cabazitaxel at a starting dose of 25 mg/m(2) intravenously over 1 h, following premedication as accepted with cabazitaxel. Treatment cycles are every 3 weeks. All patients will receive primary GCSF support.

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for this study are 18 years and older.
* Histological or cytological diagnosis of urothelial carcinoma. Mixed histologies are permitted as long as transitional cell carcinoma is the major component (i.e. > 50% of the pathologic specimen). Pure or predominant squamous cell carcinomas are not permitted.
* Patients with transitional cell carcinomas of the renal pelvis and ureter are permitted.
* Patients must have metastatic or locally advanced unresectable disease.
* Patients must have received one and only one prior chemotherapeutic regimen which included platinum (at least one cycle) for metastatic/recurrent disease. Neoadjuvant or adjuvant chemotherapy will be considered to have been first line if the patient progressed within 12 months of the last dose.
* Patients with disease progression more than 12 months following platinum based chemotherapy can be included (rather than platinum re-challenge), according to the investigator's judgment.
* ECOG performance status ≤ 2
* Estimated life expectancy of > 12 weeks.
* Patients must have measurable disease according to RECIST1.1 criteria.
* If female of childbearing potential, pregnancy test is negative within 8 days priors to first dose of study drug.
* If fertile, patient agrees to use an effective method of contraception to avoid pregnancy for the duration of the study.
* Adequate organ function; Absolute neutrophil count ≥1.5 x 109/L. Platelet count ≥ 100 x109/L. Hemoglobin ≥ 9 g/dL. Total bilirubin ≤1.0x upper limit of normal. AST/SGOT and/or ALT/SGPT ≤ 2.5x upper limit of normal. Calculated creatinine clearance > 40 ml/min (creatinine clearance will be calculated according to CKD-EPI formula: http://www.qxmd.com/calculate-online/nephrology/ckd-epi-egfr).(27)
* Able to give informed consent.

Exclusion Criteria:

* Prior taxane therapy.
* Pregnant or lactating females
* Uncontrolled brain or leptomeningeal involvement (treated brain metastasis permitted if both known lesions and medications e.g. steroids for that indication are stable).
* History of serious or concurrent illness that might be aggravated by study treatment.
* Known human immunodeficiency virus (HIV) infection or active hepatitis B/C.
* History of class II-IV congestive heart failure.
* Significant renal impairment.
* Uncontrolled hematuria.
* History of severe hypersensitivity reaction (≥grade 3) to docetaxel.
* History of severe hypersensitivity reaction (≥grade 3) to polysorbate 80 containing drugs.
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a one week wash-out period is necessary for patients who are already on these treatments) (see Appendix).
* Other malignancies except adequately controlled basal cell carcinoma of the skin or carcinoma in situ of the cervix or incidental prostate cancer (T1a, Gleason < 7 PSA < 10ng/ml) or any other tumor within 2 years prior to enrollment.
* Other investigational therapy or radiation therapy within 30 days before registration.
* Patients not willing to employ adequate contraception for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Response rate | up to 2 years
  The primary end point is objective response rate (ORR): CR+ PR, assessed according to response evaluation criteria in solid tumors (RECIST 1.1) guidelines.

SECONDARY OUTCOMES:
Clinical benefit | up to 2 years
  Secondary endpoints include clinical benefit with the following parameters: PR+CR+SD.
Duration of response | up to 2 years
  Assessment of duration of response to treatment with Cabazitaxel.
Disease control rate | up to 2 years
  Assessment of stable disease ≥ 16 weeks, PR or CR.
PFS | up to 2 years
  To determine the progression free survival (PFS) of study population defined as a 20% increase in the largest diameter of the largest lesion by CT scan.
Overall Survival | up to 2 years
  To determine the percentage of patients alive at data cutoff from trial entry. Overall survival will be measured from date of randomization to date of death due to any cause.
Safety and tolerability of treatment | up to 2 years
  Number of participants with adverse events as a measure of safety and tolerability, assessment of dose modifications according to patient's toxicity levels.
Surrogate markers to cabazitaxel | up to 3 years
  Assessment of surrogate markers to cabazitaxel response.

CONTACTS AND LOCATIONS:
Overall Officials: Avivit - Pe'er, Dr., Principal Investigator — Rambam MC
Locations (2):
- Israel (2):
  - Rambam MC, Haifa
  - Rabin Medical Center, Petah Tikva